CLINICAL TRIAL: NCT02746354
Title: Effects of a Patient Driven Assessment Process With Complex Pain Patients (PDAP)
Brief Title: Effects of a Patient Driven Assessment Process With Complex Pain Patients
Acronym: PDAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00003197
Record Dates: First submitted 2016-04-14; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Analgesics, Opioid; Primary Health Care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The MySupport tool (Experimental): Utilization of the MySupport tool, a tailored patient-centered assessment
  Interventions: Other: The MySupport tool
- Usual care (No Intervention)

INTERVENTIONS:
Other: The MySupport tool — Utilization of the MySupport tool, a tailored patient-centered assessment
  Arms: The MySupport tool

SUMMARY:
The objective of this study is to engage patients with chronic pain and other key stakeholders in an iterative process of pilot-testing a validated patient generated instrument, the Measure Yourself Medical Outcome Profile (MYMOP), to support primary care encounters and provide a direct comparison between a strategy of incorporating patient reported outcomes into the package of care for complex pain patients and usual care. The specific aims of this phase of the project are to: 1) adapt the MYMOP for use in the primary care setting well-integrated into everyday practice flow, and 2) evaluate whether the utilization of the MYMOP data in routine primary care encounters results in improvements in patient symptoms and functioning over time as well as increased satisfaction with the visit for patients and primary care providers. To achieve Aim 2, the investigators will compare the reported outcomes and health care utilization from participating patients in this study for whom the MYMOP-based instrument will be used in routine clinical care to a matched group of chronic pain patients who will not receive the MYMOP-based assessment but will otherwise have similarly collected data. This also allows us to evaluate of the extent to which use of the tool adds patient-centered information to more conventional instruments. In addition to these two aims, for a third aim, the investigators plan to collect qualitative data from patients, their family members, Kaiser Permanente Northwest (KPNW) health care providers, and KPNW administrators to better understand the needs of this subpopulation of patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Kaiser Permanente Northwest health plan members with at least 12 months of continuous eligibility at time of study entry and receive primary care from participating physicians
* Continued opioid use during the previous 6 months, as defined by 2 or more dispenses of long-acting opioids and/or a minimum cumulative supply of 90 days' worth of short-acting opioids based on electronic medical record (EMR) d) EMR recorded diagnosis of nonspecific chronic pain, Fibromyalgia, or diagnosis of ≥ 2 types of pain in the past year

Exclusion Criteria:

* Active cancer
* Substance abuse or dependence
* Hospice care
* Severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain severity and functioning | Change at 5 months, change from 5 to10 months and change at 10 months
  Brief Pain Inventory (BPI-SF): pain severity and pain interference subscales

SECONDARY OUTCOMES:
Quality of sleep | Change at 5 months, change from 5 to10 months and change at 10 months
  Insomnia Severity Index
Patient skill in managing health care | Change at 5 months, change from 5 to10 months and change at 10 months
  Patient Activation Measure
Health-related quality of life | Change at 5 months, change from 5 to10 months and change at 10 months
  EuroQuol Instrument
Clinician empathy | Change at 5 months, change from 5 to10 months and change at 10 months
  CARE measure
Self-care practices | Change at 5 months, change from 5 to10 months and change at 10 months
  Questionnaire
Health services utilization | Change at 5 months, change from 5 to10 months and change at 10 months
  Electronic medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No